CLINICAL TRIAL: NCT00269789
Title: Comparative Crossover Study of OROS (Methylphenidate HCl), Ritalin, and Placebo in Children With ADHD
Brief Title: A Comparative Effectiveness Study Evaluating OROS Methylphenidate HCl, Ritalin (Methylphenidate HCl), and Placebo for the Treatment of Attention Deficit Hyperactivity Disorder in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR005992
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; OROS®; Ritalin®; children; methylphenidate; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

ARMS (3):
- 001 (Experimental): OROS Methylphenidate HCl
  Interventions: Drug: OROS Methylphenidate HCl
- 002 (Active Comparator): Ritalin
  Interventions: Drug: Ritalin
- 003 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritalin
  Arms: 002
Drug: OROS Methylphenidate HCl
  Arms: 001
Drug: Placebo
  Arms: 003

SUMMARY:
The purpose of this study is to compare the effectiveness (onset of effect, time to loss of effect, and overall efficacy) of methylphenidate given as an OROSÂ® (methylphenidate HCl) formulation, compared to immediate-release RitalinÂ® and placebo for the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in children using standardized attention and behavior scales, and other assessments. Both OROSÂ® Methylphenidate HCl and RitalinÂ® contain the central nervous system stimulant, methylphenidate HCl.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) represents the most common neurobehavioral disorder in children, affecting 3% to 5% of the school-age population. This is a double-blind, double-dummy, randomized, placebo-controlled, active-controlled, crossover trial in children with ADHD, to compare the safety and effectiveness (onset of effect, time to loss of effect and overall efficacy) of OROS® Methylphenidate HCl with standard immediate-release Ritalin® and placebo. During this study, patients receive each of the three treatments (OROS® Methylphenidate HCl 18, 36 or 54 milligrams per day, Ritalin® 5, 10 or 15 milligrams three times per day, or placebo) for 7 days, and are assigned to one of three dosage levels depending upon their prestudy methylphenidate dose and regimen. The total study participation for each patient will be 21 days. Since ADHD is manifested in a variety of settings and can affect attention and behavior, this study assesses efficacy in home, community school, and laboratory school settings using numerous assessments designed to evaluate various aspects of the disorder. These assessments are completed by a variety of raters, including the parents/caregivers, community school teachers, laboratory school teachers and the laboratory school counselor. The primary measure of effectiveness is the community school teacher's rating on the IOWA Conners Inattention/Overactivity subscale. Additional measures of effectiveness include IOWA Conners (Inattention/Overactivity and Oppositional/Defiance subscale) ratings, SKAMP attention and deportment ratings, peer interaction and other behavioral ratings, global assessments, accuracy and productivity of independent assigned academic seatwork, and assessments of positive and negative social behaviors, classroom rule violations and disruptive behaviors. Safety evaluations include the incidence of adverse events, vital signs, sleep quality, appetite, and the presence/severity of tics (hard-to-control, repeated twitching of any parts of the body or hard-to-control repeating of sounds or words). Patients will be given oral doses of: OROS® (methylphenidate HCl) either 1, 2 or 3 of the 18 milligram tablets once daily, Ritalin® 5, 10, or 15 mg (encapsulated/single capsule) three times per day, or placebo. There are three treatment groups, each group dosing for 7 days for a total of 21 days on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of one of the three subtypes of Attention Deficit Hyperactivity Disorder (ADHD) verified by both a parent/child interview and a teacher assessment using SNAP-IV questionnaires
* taking 5 - 20 mg of immediate-release methylphenidate (Ritalin®) at least twice a day, 20 - 60 mg of sustained-release methylphenidate (Ritalin-SR®) per day, or a combination of immediate-release and sustained-release methylphenidate up to a daily dose not exceeding 60 mg
* having used methylphenidate for at least 3 months at some time in the past and have been on the same dose for the previous 4-week period without any significant adverse experiences, considered to be positive responders to methylphenidate therapy, and agreeing to take only the supplied study drug as treatment for ADHD during the three-week treatment phase of the study
* able to comply with the study visit schedule and whose parent(s) and teacher are willing and able to complete the protocol-specified assessments, including behavior modification procedures
* agreeing not to ingest any caffeine containing beverages (e.g., coffee or soda) or foods (e.g., chocolate) on days 7, 14, and 21 of the study

Exclusion Criteria:

* Patients having clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract
* considered markedly anxious, tense, agitated, or depressed, having psychotic disorders, a history of seizures, or having a diagnosis of Tourette's syndrome
* whose primary treatment focus is oppositional-defiant disorder, conduct disorder, or tics, or whose primary treatment focus is other psychiatric conditions such as depressive disorders, bipolar disorders, or other mood disorders
* having a mean of two blood pressure measurements (systolic or diastolic) equal to or greater than the 95th percentile for age, sex, and height
* if female, have begun menstruation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-03; Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
IOWA Conners Inattention/Overactivity subscale ratings by the Community School Teacher on Days 6, 13 and 20, evaluating study days 2 - 6, 9 - 13, and 16 - 20, respectively.

SECONDARY OUTCOMES:
IOWA Conners Inattention/Overactivity and Oppositional/Defiance subscale ratings; SKAMP attention and deportment ratings; Global assessments; Accuracy and completion on assigned academic tasks; Peer interactions ratings; Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Pelham WE, Gnagy EM, Burrows-Maclean L, Williams A, Fabiano GA, Morrisey SM, Chronis AM, Forehand GL, Nguyen CA, Hoffman MT, Lock TM, Fielbelkorn K, Coles EK, Panahon CJ, Steiner RL, Meichenbaum DL, Onyango AN, Morse GD. Once-a-day Concerta methylphenidate versus three-times-daily methylphenidate in laboratory and natural settings. Pediatrics. 2001 Jun;107(6):E105. doi: 10.1542/peds.107.6.e105. PMID 11389303